CLINICAL TRIAL: NCT05350761
Title: Rare Tumors and Cancer Predisposition in Individuals and Families
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000678; 000678-C
Record Dates: First submitted 2022-04-26; First posted 2022-04-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Cancer; Hereditary Neoplasms; Genetic Predisposition to Cancer; Environment
Keywords: Cancer; Genes/Genetics; Hereditary Neoplasms; Environment; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Center Cohort: includes Proband, Other carriers in family, Family Controls
- Field Cohort: includes Proband, Other carriers in family, Family Controls

SUMMARY:
Background:

Some people may be prone to develop cancer for many reasons. Factors that affect their risk include the genes they inherit and the environment they live and work in. Researchers want to learn more about the natural history of cancer.

Objective:

To understand how genes and environmental factors can cause tumors and related conditions.

Eligibility:

People of any age who:

Have tumors of an unusual type, pattern, or number

Have a family member with a history of cancer

Have been exposed to other factors that may increase their risk of cancer

Design:

This study does not involve treatment.

Participants will answer questions about their personal and family medical history. They will give permission for researchers to see their medical records.

Participants may be invited to the NIH Clinical Center for a physical exam. They may give samples including saliva, cheek cells, blood, urine, skin, and/or hair.

Participants with cancer may give bone marrow. A needle will be used to remove a small sample of bone marrow from their hip bone.

Participants may have a biopsy of their tumor.

Participants may have other exams:

Dental

Ear, nose, and throat

Eye

Hearing

Heart function and structure

Participants with cancer may undergo more exams:

A test of how much energy their body uses when resting

A sleep study with a test that measures brain electrical activity. They will have sensors attached to their body while they sleep overnight in a lab.

Imaging scans, such as CT, MRI, a test to measure how dense their bones are (DEXA), and ultrasound.

Participants will have their genes tested. A counsellor will help them understand the results.

Participants will be followed until at least 2035.

DETAILED DESCRIPTION:
Study Description: The overall purpose of this study is to comprehensively and longitudinally evaluate the natural history of participants with rare tumors, genetic syndromes, genetic variants, and/or family history consistent with or hypothesized to contribute to predisposition to cancer(s) of interest to DCEG investigators. It will also facilitate evaluation of patients who may be candidates for other NIH Clinical Center (CC) clinical trials. These individuals and families will be evaluated and followed longitudinally to define the clinical spectrum (e.g., disease course, cancer risks, response to therapies, survival) and other phenotypic manifestations associated with rare tumors, genetic variants, and cancer predisposition syndromes.

Objectives:

1. To evaluate and define the clinical spectrum (phenotype), penetrance and natural history of disease in syndromes predisposing to cancer;
2. To evaluate the phenotypes and natural history arising from known -or suspected- pathogenic germline variants in known -or suspected cancer-susceptibility genes;
3. To evaluate potential neoplastic precursor conditions in individuals and families at risk of cancer;
4. To quantify site-specific risks of such tumors in family members;
5. To discover, map, and determine inheritance patterns and functions of cancer susceptibility genes;
6. To identify etiologically or clinically relevant changes to the somatic genome in these patients;
7. To educate and counsel study participants about cancer risk including quantitative risk assessment and communication; prevention and surveillance recommendations; early detection activities; and management recommendations, when known.
8. To facilitate and enhance enrollment in interventional clinical trials within the NCI or other Institutes.

Endpoints:

Primary Endpoint: The general goals of the research conducted under this protocol are to:

1. Discover germline cancer susceptibility genes
2. Define the natural history and clinical spectrum of disease in high risk cancer susceptibility families
3. Define potential precursor states
4. Quantify risks of cancers in family members
5. Identify differences between familial and sporadic neoplasia
6. Identify genetic determinants, environmental risk factors, gene-environment, and gene-gene interactions in high risk families
7. Characterize the somatic genome of tumors from participants.

Secondary Endpoints:

1. Define penetrance of tumors in family members
2. Create full protocols for specific tumors or syndromes based on the pilot studies conducing within this study

ELIGIBILITY:
* INCLUSION CRITERIA:

Although specific familial syndromes vary in prevalence by sex, race or ethnicity, no one is excluded from participation by sex, gender, race or ethnicity. Since families participate in studies, the sex distribution is essentially balanced, and all ages are included. Minor children below the age of assent are actively studied only when the benefits of participation outweigh the risks.

Affected: An individual who meets any of the following criteria will be eligible to participate in this study:

1. Personal medical history of neoplasia of an unusual type, pattern, or number; or,
2. Known or suspected factor(s) predisposing to neoplasia, either genetic and/or congenital factors (birth defects, metabolic phenotype, chromosomal anomalies or Mendelian traits associated with tumors), environmental exposure (medications, occupation, radiation,

   diet, infectious agents, etc.), or unusual demographic features (very young age of onset, multiple tumors, etc.).
3. There is no age restriction; therefore including viable neonates However, children < 3 years old will not come to the Clinical Center unless clinically indicated until they are >= 3 years old.
4. Participant or their Legally Authorized Representative (LAR) must sign and date an IRB approved informed consent form (signed on paper or electronically for the Field Cohort / signed on paper for the Clinic Center Cohort)

Unaffected Controls: An individual who meets any of the following criteria will be eligible to participate in this study:

1. Family medical history of neoplasia of an unusual type, pattern, or number; or,
2. Known or suspected factor(s) predisposing to neoplasia, either genetic and/or congenital factors (birth defects, metabolic phenotype, chromosomal anomalies or Mendelian traits associated with tumors), environmental exposure (medications, occupation, radiation,

   diet, infectious agents, etc.), or unusual demographic features (very young age of onset, multiple tumors, etc.).
3. There is no age restriction; therefore including viable neonates. However, children < 3 years old will not come to the Clinical Center unless clinically indicated until they are >= 3 years old.
4. Participant or their LAR must sign and date an IRB-approved informed consent form (signed on paper or electronically for the Field Cohort / signed on paper for the Clinic Center Cohort)

Personal and family medical history will be verified through questionnaires, interviews, and review of pathology slides and medical records. For familial neoplasms, two or more living affected cases among family members are required. The types of suspected factors predisposing to neoplasia and/or familial tumors under active accrual and study will be investigator- and hypothesis-driven. This approach permits CGB investigators to remain alert to the opportunities afforded by clusters of rare tumors in families and individuals, and to be more responsive to the dynamic research priorities in cancer genetics.

EXCLUSION CRITERIA:

Affected: An individual who meets any of the following criteria will be excluded from participation in this study:

1. Referred individuals for whom reported diagnoses cannot be verified
2. Inability of the participant or LAR to understand and be willing to sign a written informed consent document.
3. Referred individuals who are eligible for other CGB protocols that are specific to a hereditary cancer syndrome (e.g., Li-Fraumeni Syndrome, Familial Melanoma) Unaffected Controls: An individual who meets any of the following criteria will be excluded

from participation in this study:

1. Referred families for whom reported diagnoses cannot be verified
2. Inability of the participant or LAR to understand and be willing to sign a written informed consent document.
3. Referred families who are eligible for other CGB protocols that are specific to a hereditary cancer syndrome (e.g., Li-Fraumeni Syndrome, Familial Melanoma)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical; volunteers come from all across the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Defining the natural history of familial cancers and susceptibility states over multiple generations, identifying cancer susceptibility genes, and assessing gene-environment and gene-gene interactions | Ongoing
  New cancer development or current health status

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Savage, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NIH National Cancer Institute - Shady Grove, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Genotype and sequence data along with clinical phenotypes will be deposited in a genomic database in accordance with current NIH Genomic Data Sharing (GDS) Policy and the NIH Human Data Sharing Policy.@@@@@@The following human data generated in this research will be shared for future research as follows:@@@@@@De-identified data in an NIH-funded or approved public repository.@@@@@@De-identified data in BTRIS (automatic for activities in the Clinical Center)@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements.@@@@@@The data will be shared at the time of publication or shortly after.@@@@@@Unlinked genomic data will be deposited in public genomic databases such as dbGaP in compliance with the NIH Genomic Data Sharing Policy.
Supporting Information: SAP, ICF
Time Frame: The data will be shared at the time of publication or shortly after.
Access Criteria: Section 9.10 titled Publication and Data Sharing Policy in the protocol which describes the plan for data sharing plans including human data sharing and genomic data sharing.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000678-C.html